CLINICAL TRIAL: NCT05277259
Title: Comparative Effects of Conventional Physical Therapy, Kinesio Taping and Extracorporeal Shock Wave Therapies in Upper Trapezius Myofascial Pain Syndrome.
Brief Title: Comparative Effects of Conventional Physical Therapy, Kinesio Taping and ESWT in Upper Trapezius MPS.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Volkan Şah, Principal Investigator, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: van yyü university
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Trapezius Muscle Strain
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Extracorporeal Shock Wave Therapy (Active Comparator): Extracorporeal shock wave therapy (ESWT) is a noninvasive treatment that involves delivery of shock waves to injured soft tissue to reduce pain and promote healing.
  Interventions: Device: Extracorporeal Shock Wave Therapy
- Kinesiotaping (Active Comparator): The Kinesiotaping method is a therapeutic taping technique which alleviates pain.
  Interventions: Other: Kinesiotaping
- Conventional Physical Therapy (Active Comparator): Hotpack, therapeutic ultrasound and tens applications.
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Device: Extracorporeal Shock Wave Therapy — Device named 'Elettronica Pagani,Italy' and will be used with radial probe.
  Arms: Extracorporeal Shock Wave Therapy
Other: Kinesiotaping — Elastic band to be used to stretch the upper trapezius muscle in the desired direction.
  Arms: Kinesiotaping
Other: Conventional Physical Therapy — Conventional physical therapy will be consisted of hotpack, therapeutic ultrasound and tens applications.
  Arms: Conventional Physical Therapy

SUMMARY:
There is no study in the literature comparing both kinesiotaping and Extracorporeal Shock Wave Therapy (ESWT) with conventional physical therapy in upper trapezius myofascial pain syndrome. In this study, we aimed to make this comparison.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least 1 active trigger point in the upper trapezius muscle, exacerbation of pain when this point(s) is pressed, painful limitation of cervical lateral flexion and extension.

Exclusion Criteria:

* Having a history of spine and upper extremity surgery, neuromuscular disease, active rheumatologic disease, active infection, malignancy, having previously applied ESWT or Kinesio Taping to the back and neck region.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | at baseline (before the treatment)
  patient's self-assessment of pain, in the range of 0 to 10, higher scores mean a worse outcome.
Visual Analogue Scale (VAS) | 2 weeks after baseline (at the end of treatment)
  patient's self-assessment of pain, in the range of 0 to 10, higher scores mean a worse outcome
Visual Analogue Scale (VAS) | 6 weeks after baseline (one month after the end of treatment)
  patient's self-assessment of pain, in the range of 0 to 10, higher scores mean a worse outcome
Neck Disability Index (NDI) | at baseline (before the treatment)
  a self-report questionnaire used to determine how neck pain affects a patient's daily life and to assess the self-rated disability of patients with neck pain. The total score ranges from 0 (no disability) to 50 (total disability).
Neck Disability Index (NDI) | 2 weeks after baseline (at the end of treatment)
  a self-report questionnaire used to determine how neck pain affects a patient's daily life and to assess the self-rated disability of patients with neck pain. The total score ranges from 0 (no disability) to 50 (total disability).
Neck Disability Index (NDI) | 6 weeks after baseline (one month after the end of treatment)
  a self-report questionnaire used to determine how neck pain affects a patient's daily life and to assess the self-rated disability of patients with neck pain. The total score ranges from 0 (no disability) to 50 (total disability).

SECONDARY OUTCOMES:
Measurement of Cervical range of motion (Cervikal ROM) | at baseline (before the treatment)
  Measuring cervical lateral flexion and cervical extension with a manual goniometer.
Measurement of Cervical range of motion (Cervikal ROM) | 2 weeks after baseline (at the end of treatment).
  Measuring cervical lateral flexion and cervical extension with a manual goniometer.
Measurement of Cervical range of motion (Cervikal ROM) | 6 weeks after baseline (one month after the end of treatment)
  Measuring cervical lateral flexion and cervical extension with a manual goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Volkan Şah, Principal Investigator — Yüzüncü Yıl Üniversitesi Tıp Fakültesi
Locations (1):
- Yuzuncu Yil University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No